CLINICAL TRIAL: NCT01732471
Title: A Phase III Non-comparative Open-label Clinical Study to Evaluate the Response to and Safety of Kuvan (Sapropterin Dihydrochloride) After 6 Weeks of Treatment in Patients of 4 to 18 Years of Age With Phenylketonuria Who Have Elevated Blood Phenylalanine Levels
Brief Title: Phase 3 Open-label Study to Evaluate the Response and Safety of Kuvan® in Subjects With Phenylketonuria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR 700773_510
Record Dates: First submitted 2012-11-19; First posted 2012-11-22 (Estimated); Results first posted 2014-07-28 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Phenylketonuria
Keywords: EMR 700733_510, Genetic disorder, Phenylketonuria, phenylalanine, Kuvan, sapropterin dihydrochloride
MeSH Terms: conditions — Phenylketonurias; Genetic Diseases, Inborn | interventions — sapropterin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Kuvan® (Experimental)
  Interventions: Drug: Kuvan®

INTERVENTIONS:
Drug: Kuvan® — Kuvan® (sapropterin dihydrochloride) will be administered orally at a dose of 20 milligram per kilogram per day (mg/kg/day) once daily for 8 days. If there is 30 percent (%) decrease in blood phenylalanine levels from baseline at the end of Day 8, then treatment will be continued at the same dose for further 6 weeks.
  Other Names: Sapropterin dihydrochloride; 6R-BH4 tetrahydrobiopterin

SUMMARY:
This is an open-label, non-comparative, Phase 3 study to evaluate the degree, frequency of response and safety of Kuvan® (sapropterin dihydrochloride) in subjects aged 4 to 18 years who have phenylketonuria and with elevated blood phenylalanine level of greater than or equal to 450 micromole per liter.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent (for children under 18 years old the parent[s]/guardians give informed consent, subjects 14-17 years old give additionally their own written informed consent)
* Age of 4 - 18 years, inclusive
* Confirmed clinical and biochemical hyperphenylalaninemia due to phenylketonuria documented by past medical history with at least 2 blood phenylalanine level greater than or equal to 400 micromole per liter obtained in 2 separate occasions
* Blood phenylalanine level at screening greater than or equal to 450 micromole per liter (mean of two measurements)
* For women of childbearing potential, a negative urine pregnancy test is required at screening and willingness to use a highly effective method of contraception is required while participating in the study
* Subject and/or the parent/guardian willing and able to comply with study procedures
* Subject and/or the parent/guardian willing to continue current diet unchanged during the 8 days response test and to adapt the diet according to phenylalanine therapeutic target range during the 6 week treatment period

Exclusion Criteria:

* Subject already assessed for responsiveness to sapropterin dihydrochloride or other tetrahydrobiopterin (BH4)
* Used any investigational agent other than Kuvan® (sapropterin dihydrochloride) within 30 days of screening, or required any investigational agent or vaccine prior to completion of all scheduled study assessments
* Pregnant or breastfeeding, or considering pregnancy
* Concurrent disease or conditions that would interfere with study participation or safety (for example, seizure disorder, asthma or other condition requiring oral or parenteral corticosteroid administration, insulin-dependent diabetes, or organ transplantation recipient)
* Concurrent use of required concomitant treatment with any drug known to inhibit folate synthesis (for example, methotrexate), levodopa, phosphodiesterase type-5 (PDE-5) inhibitors (such as, sildenafil, vardenafil or tadalafil), medications that are known to affect nitric oxide synthesis metabolism or action
* Any conditions, that, in the view of the Principal Investigator renders the subject at high risk for failure to comply with treatment or to complete the study
* Clinical diagnosis of primary BH4 deficiency
* Known hypersensitivity to Kuvan® (sapropterin dihydrochloride) or its excipients or to other approved or non-approved formulation of tetrabiopterin

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2012-11; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Please contact Merck KGaA Communication Center, Darmstadt, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Kuvan®: Kuvan® (sapropterin dihydrochloride) was administered orally at a dose of 20 milligram per kilogram per day (mg/kg/day) once daily for 8 days. If there is 30 percent (%) decrease in blood phenylalanine levels from baseline at the end of Day 8, then treatment was continued at the same dose for further 6 weeks.
Period: Overall Study
Arm/Group | Kuvan®
Started | 90
Completed | 89
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Intention to Treat (ITT) population included all participants who had efficacy assessment result from at least 1 visit except for the inclusion visit.
Groups:
- Kuvan®: Kuvan® (sapropterin dihydrochloride) was administered orally at a dose of 20 mg/kg/day once daily for 8 days. If there is 30 percent (%) decrease in blood phenylalanine levels from baseline at the end of Day 8, then treatment was continued at the same dose for further 6 weeks.
Arm/Group | Kuvan®
Number analyzed (Participants) | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.59 (4.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 49

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Response to Kuvan® (Sapropterin Dihydrochloride) Treatment
Description: Response to Kuvan® (sapropterin dihydrochloride) treatment was defined as a reduction in blood phenylalanine levels of greater than or equal to 30% at Day 8 as compared to baseline.
Time Frame: Day 8
Population: Overall (ITT) population included all participants who had efficacy assessment result from at least 1 visit except for the inclusion visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Kuvan®
Number analyzed (Participants) | 90
percentage of participants | 33.3 [23.7 to 44.1]

2. Secondary Outcome: Percent Change From Baseline in Blood Phenylalanine Levels at Day 8 in Overall Population
Description: Percent change in blood phenylalanine levels after 8-day Kuvan® therapy (response test period) was calculated as (blood phenylalanine level at Day 8 minus blood phenylalanine level at baseline)*100/ blood phenylalanine level at baseline.
Time Frame: Baseline, Day 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Kuvan®
Number analyzed (Participants) | 90
percent change | -14.14 (28.35)

3. Secondary Outcome: Percent Change From Baseline in Blood Phenylalanine Levels at Day 8 in Sub-population of Responders
Description: as for outcome 2
Time Frame: Baseline, Day 8
Population: Sub-population of responders included participants with reduction in blood phenylalanine levels of greater than or equal to 30% at Day 8 as compared to baseline.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Kuvan®
Number analyzed (Participants) | 30
percent change | -44.25 (15.13)

4. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) in Overall Safety Population
Description: An adverse event (AE) was defined as any new untoward medical occurrences/worsening of pre-existing medical condition without regard to possibility of causal relationship. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect.
Time Frame: Baseline up to Week 11
Population: Overall safety population included all participants who received at least 1 dose of investigational medicinal product.
Measure: Number; unit: participants
Arm/Group | Kuvan®
Number analyzed (Participants) | 90
participants
  AEs | 24
  SAEs | 1

ADVERSE EVENTS:
Time Frame: Baseline up to Week 11
Description: An AE is any new untoward medical occurrences/worsening of pre-existing medical condition without regard to possibility of causal relationship. An SAE is an AE resulting in any of following outcomes:death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect.
Arm/Group | Kuvan®
Serious Adverse Events (participants affected / at risk) | 1/90
Other Adverse Events (participants affected / at risk) | 23/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Kuvan® (N=90)
Upper limb fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Kuvan® (N=90)
Anaemia (Blood and lymphatic system disorders) | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1
Faeces pale (Gastrointestinal disorders) | 1
Gastroduodenitis (Gastrointestinal disorders) | 1
Genital labial adhesions (Reproductive system and breast disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Heat stroke (Injury, poisoning and procedural complications) | 1
Iodine deficiency (Metabolism and nutrition disorders) | 1
Leukocyturia (Renal and urinary disorders) | 1
Myopia (Eye disorders) | 1
Oral herpes (Infections and infestations) | 1
Phenylketonuria (Renal and urinary disorders) | 2
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory tract infection viral (Respiratory, thoracic and mediastinal disorders) | 9
Retinal vascular disorder (Vascular disorders) | 2
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 1
Syncope (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All written or oral publications and/or information related to Study and/or results of Study should be submitted at first in writing to Sponsor at least 30 working days for publication and 15 working days for brief review, abstract before planned date of submission. If Sponsor is filing a patent application on Study results, Sponsor can delay its authorization for publication/communication of Study results to Investigator and/or Research Centre until date of international registration of patent.